CLINICAL TRIAL: NCT06417203
Title: Hypobaric Spinal or Hyperbaric in Partial Hip Arthroplasty Surgeries? Can an Answer be Found by Perfusion Index?
Brief Title: Hypobaric Spinal or Hyperbaric in Partial Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, Associate Professor,MD, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11.05.2024-ADYU-ANS-NY-05
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: two gropus planned for study
  1. group - Hyperbaric spinal anesthesia
  2. group - Hypobaric spinal anesthesia
Who Masked: Participant, Outcomes Assessor
Masking Description: for patient - closed envelope system for Outcomes Assessor - will not participate perioperative period and will not know group of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyberbaric group (Experimental): In this group, hyperbaric bupivacaine was planned to use in spinal anesthesia for partial hip replacement surgery
  Interventions: Procedure: spinal anesthesia with hyberbaric bupivacaine
- Hypobaric group (Experimental): In this group, hypobaric bupivacaine was planned to use in spinal anesthesia for partial hip replacement surgery
  Interventions: Procedure: spinal anesthesia with hypobaric bupivacaine

INTERVENTIONS:
Procedure: spinal anesthesia with hyberbaric bupivacaine — After standard ASA monitoring in the operation room, spinal anaesthesia was induced by injection of 10 mg hyperbaric bupivacaine into the subarachnoid space with the help of a spinal needle through the L4-5 intervertebral space. (modified from the initially registered 12.5 mg due to the higher incidence of hypotension and bradycardia observed with 12.5 mg in our institutional practice, prompting a safety-driven revision)
  Arms: Hyberbaric group
Procedure: spinal anesthesia with hypobaric bupivacaine — After standard ASA monitoring in the operation room, spinal anaesthesia was induced by injection of 10 mg hypobaric bupivacaine into the subarachnoid space with the help of a spinal needle through the L4-5 intervertebral space. (modified from the initially registered 12.5 mg due to the higher incidence of hypotension and bradycardia observed with 12.5 mg in our institutional practice, prompting a safety-driven revision)
  Arms: Hypobaric group

SUMMARY:
The aim of this study was to compare the effects of hypobaric and hyperbaric spinal applications on patient haemodynamics, duration of anaesthetic effect and postoperative analgesia. Thus, it was aimed to determine the method that protects haemodynamics more and suppresses postoperative pain complaints of patients better in this patient group with advanced age, comorbid systemic diseases and high risk of operation.

DETAILED DESCRIPTION:
Patients who are planned to be operated for partial hip replacement at Adıyaman University Training and Research Hospital, who are informed about the study and who agree to participate in the study with their written consent will be included in the study.

Patients who agree to participate in the study will be divided into two groups: hypobaric and hyperbaric spinal anaesthesia patients will be divided into two groups to be decided by the Anaesthesiology and Reanimation specialist responsible for the operation (hyperbaric/hypobaric). Before the start of the operation, perfusion index (PI) values will be monitored with a probe in both lower extremities with standard ASA monitoring. Haemodynamic values (blood pressure arterial, peak heart rate, peripheral oxygen saturation), PI values of both extremities, duration of motor and sensory block, postoperative numeric pain scores of all patients will be recorded and these values will be compared in both groups.

Thus, it was aimed to compare the efficacy, safety, block times and contribution to pain management of each application.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* 18-65 aged

Exclusion Criteria:

* ASA III-IV
* Deny to participiate
* conditions that spinal anesthesia contraindicated
* use of alpha or beta-blockers
* allergy to local anesthetics
* diabetes mellitus
* peripheral vascular disease (The following exclusion criteria were added to ensure patient safety and to avoid confounding factors that could interfere with perfusion index measurements or hemodynamic responses: use of alpha or beta-blockers, diabetes mellitus, and peripheral vascular disease. These conditions may significantly alter autonomic regulation, vascular tone, or peripheral circulation, potentially affecting perfusion index values or increasing the risk of adverse reactions to spinal anesthesia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Visual analog pain score (VAS) | First postoperative 24 hours (The originally registered follow-up period of 3 months was entered in error. The intended and actual outcome assessment period for this study is the first 24 postoperative hours.)
  a tool that asses patinet paiin level 0 (no pain) -10 (the worst pain ever had) , the tool will be used at postopertaive period

SECONDARY OUTCOMES:
Quality of recovery (QoR-15) | first postoperative24 hours(The originally registered follow-up period of 3 months was entered in error. The intended and actual outcome assessment period for this study is the first 24 postoperative hours, as correctly stated in the description section)
  a tool that asses recovery quality of patient with 15 question will be used 24th hour after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman Training and Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided